CLINICAL TRIAL: NCT07312461
Title: Causes and Management of Children Presenting With Macroscopic Hematuria in the Pediatric Emergency Department
Acronym: HMUP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9456
Record Dates: First submitted 2025-12-10; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Macroscopic Hematuria
Keywords: Macroscopic hematuria; Hematuria in children

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Macroscopic hematuria. is a common symptom, leading to numerous emergency department visits in children of all ages.

It can be linked to many pathologies, and its management in the emergency department is not standardized.

Few articles describe the management of this symptom during pediatric emergency department visits.

Therefore, it is important to study this symptom and its management in order to establish a protocol.

ELIGIBILITY:
Inclusion Criteria:

* Minor subject (<18 years old)
* Patient presenting to the pediatric emergency department with gross hematuria

Exclusion Criteria:

- Subject (and/or their parents) who expressed their opposition to participating in the study.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minor subject (<18 years old) presenting to the pediatric emergency department with gross hematuria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Describe the different causes of this symptom | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pédiatrie 1 - Réanimation - CHU de Strasbourg - France, Strasbourg, France